CLINICAL TRIAL: NCT02242617
Title: Adherence and Preference of Continuous Positive Airway Pressure Versus Mandibular Advancement Splints in Obstructive Sleep Apnea Patients: A Randomized Trial
Acronym: CHOICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Université de Montréal (Other); Laval University (Other)
Responsible Party: Principal Investigator, Fernanda Almeida, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H14-01215; RN325361 (Other Grant/Funding Number: Canadian Institute of Health Research (CIHR))
Record Dates: First submitted 2014-08-29; First posted 2014-09-17 (Estimated); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: Adherence; CPAP; Oral Appliance; Mandibular Advancement Splints; Preference
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure; Occlusal Splints

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MAS-PAP (Active Comparator): Mandibular advancement splints (MAS): dental splints used to keep the mandible in an advanced position opening the upper airway during sleep; followed by positive airway pressure (PAP)
  Interventions: Device: Positive Airway Pressure (PAP); Device: Mandibular Advancement Splints (MAS)
- PAP-MAS (Active Comparator): Positive airway pressure (PAP): a device which consists of a face mask attached to a plastic tube and a machine that blows compressed air through a patient's airway during sleep to keep the airway open; followed by mandibular advancement splints (MAS)
  Interventions: Device: Positive Airway Pressure (PAP); Device: Mandibular Advancement Splints (MAS)

INTERVENTIONS:
Device: Positive Airway Pressure (PAP) — Continuous or auto-adjusting positive airway pressure (i.e. CPAP, APAP, and described here as PAP): a device which consists of a face mask attached to a plastic tube and a machine that blows compressed air through a patient's airway during sleep to keep the airway open
  Other Names: CPAP, auto-CPAP, APAP
Device: Mandibular Advancement Splints (MAS) — Mandibular advancement splints (MAS): dental splints used to keep the mandible in an advanced position opening the upper airway during sleep
  Other Names: Oral appliance; Mandibular advancement devices; Somnodent device

SUMMARY:
Obstructive sleep apnea (OSA) is a major health problem affecting over 1,000,000 Canadians. It is the cause of significant healthcare costs with increased morbidity and mortality. The two most common and effective therapies used to treat OSA are: (1) Continuous or Automatic Positive Airway Pressure (PAP), and (2) Mandibular Advancement Splints (MAS). While both therapies reduce upper airway collapse during sleep, they differ in efficacy, acceptance, cost and side-effects, but surprisingly are similar in improving quality of life, sleepiness and blood pressure. PAP is more effective in reducing apneas while MAS is easier to use. Until now, studies have used self-reported adherence data on MAS versus objective adherence on PAP. Many studies have hypothesized that the sub-optimal efficacy with MAS therapy is counterbalanced by the superior adherence relative to PAP, resulting in a similar effectiveness for both treatments. Compliance smart chips are a recent innovation for MAS and could be used to prove this hypothesis and allow a new and complete comparison of effectiveness (efficacy + adherence) between MAS and PAP. Understanding the patient's objective adherence and long-term symptomatic improvement would provide vital information to doctors and dentists in choosing the right treatment for patients. Sixty OSA patients will receive both PAP and MAS in a random sequence. This innovative study lead by two experienced new investigators, and a research team of multidisciplinary experts, will assess objective adherence, treatment efficacy, patient preference, sleepiness and quality of life of each treatment used at home for 1 month per treatment. After this, patients will be able to go back and forth between both treatments during an additional 6-month period. The results of this study will be used by healthcare policy makers as well as clinicians who need to be part of the treatment plan decision for the many Canadians who suffer from sleep apnea.

DETAILED DESCRIPTION:
The primary aim of this study is to assess objective adherence to treatment, for PAP and MAS, and to evaluate if there will be similar effectiveness (efficacy+adherence) between PAP and MAS treatment for patients with mild to severe OSA. The secondary aim is to assess if patient preference does correlate to the final treatment adherence. An exploratory aim is to assess if the strategy of patients having both treatments available to use interchangeably could further improve treatment adherence, sleepiness, quality of life and fatigue. Having a better insight into patient adherence will improve the cost-effectiveness of treatment and will improve the health and quality of life for many Canadians who suffer from sleep apnea.

The proposed trial is a randomized open-label, two-treatment, two-period cross-over trial followed by an observational trial. Sixty OSA patients (10≤AHI≤50) will receive both PAP and MAS. As a recent innovation, we have adherence monitors for MAS that can give a new and comprehensive comparative analysis of the effectiveness between MAS and PAP. In the randomized trial phase the two treatments will be used separately for 1 month each (after treatment adaptation/titration of 1-2 months for each device). Treatment efficacy and daily treatment use data will be assessed together with changes in symptoms (quality of life, sleepiness and fatigue). Patient initial preference will be determined by using a patient decision aid. This will be followed by the observational trial phase, where all patients will have access to both interventions at home for 6 months and be allowed to choose on a daily basis the intervention to use. The intervention duration of 6 months is to allow for a sustained response in long-term adherence and to observe changes in quality of life.

ELIGIBILITY:
Inclusion Criteria:

You may be able to participate in this study if:

* You are naïve to treatment (never used CPAP or oral appliance, nor had surgery for sleep apnea);
* You are between 19-75 years old;
* You have a Body Mass Index (BMI) ≤ 35;
* You have enough teeth (at least 8 per arch) for MAS;
* You have:

  * an Apnea-Hypopnea Index (AHI) within the range 10 ≤ AHI ≤ 50 documented with polysomnography in the last 2 years; ***OR***
  * a Respiratory Disturbance Index (RDI) within the range 20 ≤ RDI ≤ 50 documented with level III portable sleep test; ***OR***
  * an Oxygen Desaturation Index (ODI) ≥ 10; and
* You have had a sleep test within the past 2 years.

Exclusion Criteria:

You may not be able to participate in this study if:

* You have extensive periodontal disease with significant tooth mobility (disease around your teeth);
* You are unable to protrude the jaw (unable to extend your jaw);
* You have a lack of a sufficient vertical opening to accommodate an appliance;
* You have uncontrolled congestive heart failure (defined as a prior clinical diagnosis, an ejection cutoff of 40% or a clinical sign in the opinion of a primary care physician or cardiologist) that makes it unsafe for you to participate in the trial in the opinion of the investigators;
* You have coronary artery disease unless stable for at least 6 months and considered by the investigators to have a stable disease;
* You have a history of angina (chest pain when your heart does not get enough blood), myocardial infarction (heart attack) or stroke;
* You have a history of major depressive disorder (such as bipolar disorder) along with current moderate or severe disease;
* You have cancer unless in remission (decreasing signs of your cancer being present) for more than 1 year;
* You have known renal (kidney) failure with need for dialysis;
* You are pregnant (if a female participant becomes pregnant during the trial, she will be withdrawn from the study);
* You have had a near miss or prior automobile accident due to sleepiness within the past 12 months; and/or
* At nighttime, 30% of the night is at ≤ 90% oxygen saturation levels.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Objectively measured adherence (hours/night and nights/week of intervention use). | At 1 month in the MAS treatment arm
  Measuring objective adherence (hours/night and nights/week of intervention use), indicated by the smart chips and symptoms.
Objectively measured adherence (hours/night and nights/week of intervention use). | At 1 month in CPAP treatment arm
  Measuring changes in objectively measured adherence (hours/night and nights/week of intervention use), indicated by the smart chips and symptoms.
Objectively measured adherence (hours/night and nights/week of intervention use). | At 1 month of using both treatments interchangeably.
  Measuring changes in objectively measured adherence (hours/night and nights/week of intervention use), indicated by the smart chips and symptoms.
Objectively measured adherence (hours/night and nights/week of intervention use). | At 6 months of using both treatments interchangeably
  Measuring changes in objectively measured adherence (hours/night and nights/week of intervention use), indicated by the smart chips and symptoms.

SECONDARY OUTCOMES:
Apnea-hypopnea index | At baseline
  Measuring apnea-hypopnea index (events/hour of sleep from Stardust-Phillips Respironics) to measure intervention efficacy (e.g. AHI)
Functional Outcomes of Sleep Questionnaire (FOSQ) responses | At baseline
  Measuring Functional Outcomes of Sleep Questionnaire (FOSQ) responses to evaluate disease specific quality of life.
Epworth Sleepiness Scale (ESS) questionnaire responses. | At baseline
  Measuring responses to Epworth Sleepiness Scale (ESS) Questionnaire to compare daytime sleepiness.
Chalder fatigue scale questionnaire responses | At baseline
  Measuring responses to the Chalder fatigue scale which assesses fatigue in the present state.
SF-36 survey responses | At baseline
  Measuring SF-36 survey responses which assesses general health status.
Apnea-hypopnea index | At 1 month in MAS treatment arm
  Measuring changes in apnea-hypopnea index (events/hour of sleep from Stardust-Phillips Respironics) to measure intervention efficacy (e.g. AHI)
Apnea-hypopnea index | At 1 month in CPAP treatment arm
  Measuring changes in apnea-hypopnea index (events/hour of sleep from Stardust-Phillips Respironics) to measure intervention efficacy (e.g. AHI)
Functional Outcomes of Sleep Questionnaire (FOSQ) responses. | At 1 month in MAS treatment arm
  Measuring changes in Functional Outcomes of Sleep Questionnaire (FOSQ) responses to evaluate disease specific quality of life.
Functional Outcomes of Sleep Questionnaire (FOSQ) responses. | At 1 month of using both treatments interchangeably
  Measuring changes in Functional Outcomes of Sleep Questionnaire (FOSQ) responses to evaluate disease specific quality of life.
Functional Outcomes of Sleep Questionnaire (FOSQ) responses | At 6 months of using both treatments interchangeably
  Measuring changes in Functional Outcomes of Sleep Questionnaire (FOSQ) responses to evaluate disease specific quality of life.
Functional Outcomes of Sleep Questionnaire (FOSQ) responses. | At 1 month in CPAP treatment arm
  Measuring changes in Functional Outcomes of Sleep Questionnaire (FOSQ) responses to evaluate disease specific quality of life.
Epworth Sleepiness Scale (ESS) questionnaire responses. | At 1 month in MAS treatment arm
  Measuring changes in Epworth Sleepiness Scale (ESS) Questionnaire responses to compare daytime sleepiness.
Epworth Sleepiness Scale (ESS) questionnaire responses. | At 1 month in CPAP treatment arm.
  Measuring changes in responses to Epworth Sleepiness Scale (ESS) Questionnaire to compare daytime sleepiness
Epworth Sleepiness Scale (ESS) questionnaire responses | At 1 month of using both treatments interchangeably
  Measuring changes in responses to Epworth Sleepiness Scale (ESS) Questionnaire to compare daytime sleepiness.
Epworth Sleepiness Scale (ESS) questionnaire responses. | At 6 months of using both treatments interchangeably.
  Measuring changes in responses to Epworth Sleepiness Scale (ESS) Questionnaire to compare daytime sleepiness.
Chalder fatigue scale questionnaire responses | At 1 month in MAS treatment arm
  Measuring changes in responses to the Chalder fatigue scale which assesses fatigue in the present state.
Chalder fatigue scale questionnaire responses | At 1 month in CPAP treatment arm
  Measuring changes in responses to the Chalder fatigue scale which assesses fatigue in the present state.
Chalder fatigue scale questionnaire responses | At 1 month of using both treatments interchangeably
  Measuring changes in responses to the Chalder fatigue scale which assesses fatigue in the present state.
Chalder fatigue scale questionnaire responses | At 6 months of using both treatments interchangeably.
  Measuring changes in responses to the Chalder fatigue scale which assesses fatigue in the present state.
SF-36 survey responses. | At 1 month in MAS treatment arm
  Measuring changes in SF-36 survey responses which assesses general health status.
SF-36 survey responses. | At 1 month in CPAP treatment arm.
  Measuring changes in SF-36 survey responses which assesses general health status.
SF-36 survey responses. | At 1 month of using both treatments interchangeably.
  Measuring changes in SF-36 survey responses which assesses general health status.
SF-36 survey responses. | At 6 months of using both treatments interchangeably.
  Measuring changes in SF-36 survey responses which assesses general health status.

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda R Almeida, DDS, MSc, PhD, Principal Investigator — University of British Columbia
Locations (3):
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - University of Montreal / Université de Montréal, Montreal, Quebec
  - Laval University / Université Laval, Québec

REFERENCES:
- [Background] Almeida FR, Mulgrew A, Ayas N, Tsuda H, Lowe AA, Fox N, Harrison S, Fleetham JA. Mandibular advancement splint as short-term alternative treatment in patients with obstructive sleep apnea already effectively treated with continuous positive airway pressure. J Clin Sleep Med. 2013 Apr 15;9(4):319-24. doi: 10.5664/jcsm.2576. PMID 23585745
- [Derived] Alshhrani WM, Hamoda MM, Okuno K, Kohzuka Y, Fleetham JA, Ayas NT, Comey R, Almeida FR. The efficacy of a titrated tongue-stabilizing device on obstructive sleep apnea: a quasi-experimental study. J Clin Sleep Med. 2021 Aug 1;17(8):1607-1618. doi: 10.5664/jcsm.9260. PMID 33745505